CLINICAL TRIAL: NCT01522768
Title: A Phase II Study of Afatinib and Paclitaxel in Patients With Advanced HER2-Positive Trastuzumab Refractory Advanced Esophagogastric Cancer
Brief Title: Afatinib and Paclitaxel in Patients With Advanced HER2-Positive Trastuzumab-Refractory Advanced Esophagogastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Boehringer Ingelheim (Industry); University of Southern California (Other); Dana-Farber Cancer Institute (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-166
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: ESOPHAGUS; STOMACH; Afatinib; paclitaxel; trastuzumab; 11-166
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Afatinib; Paclitaxel

ARMS (1):
- Afatinib and Paclitaxel (Experimental): This is a multi-institution, open-label, non-randomized, Phase II evaluation of oral afatinib daily and intravenous paclitaxel (weekly, 3 weeks on, 1 week off) in patients with trastuzumab refractory HER2-positive metastatic or recurrent esophagogastric adenocarcinoma. An initial biopsy prior to the start of therapy is required for the correlative studies evaluating the biologic effects of afatinib. It will be obtained for all patients whose tumors are feasible to biopsy. At the site investigator's discretion, a second biopsy will also be obtained. At the discretion of the MSK Principal Investigator, select participants who show response on this study and then progress may be asked to have an optional third biopsy.
  Interventions: Drug: Afatinib and Paclitaxel

INTERVENTIONS:
Drug: Afatinib and Paclitaxel — All patients receiving therapy on trial with afatinib and trastuzumab will continue on afatinib and trastuzumab until disease progression or intolerable toxicity. All additional patients will be enrolled on afatinib and paclitaxel. Patients will be treated with afatinib and paclitaxel combination. Patients will receive oral afatinib 40 mg daily plus paclitaxel 80 mg/m^2 intravenously on day 1, 8, and 15 of a 28-day cycle.

SUMMARY:
The purpose of this study is to find out what effects, good or bad, the combination of standard chemotherapy agent paclitaxel with the investigational (experimental) drug afatinib that targets HER2, has on HER2-positive esophagogastric cancer that started to get bigger despite previous treatment with trastuzumab. The doctors will also study the tumor to understand why it grew while on trastuzumab treatment and to see the effects afatinib and paclitaxel has on the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed esophagogastric cancer.
* HER2 overexpression and/or amplification as determined by immunohistochemistry (3+) or FISH (≥2.0)
* Previously received trastuzumab as part of a regimen in the perioperative or metastatic setting with evidence of progression 9Zr-trastuzumab use as imaging agent for 89Zr-trastuzumab PET permitted..
* May have previously received lapatinib as part of a regimen in the perioperative or metastatic setting with evidence of progression of disease. Washout period for lapatinib of 14 days.
* Completion of previous chemotherapy regimen ≥2 weeks prior to the start of study treatment. Other chemotherapy regimens may have been administered between the time of progression on prior trastuzumab containing regimen and protocol therapy. No restriction on prior chemotherapy regimens for advanced stage disease.
* At least one measurable metastatic lesion according to RECIST 1.1 criteria. Ascites, pleural effusions, and bone metastases are not considered measurable. Minimum indicator lesion size = 10 mm by helical CT or = 20 mm by conventional techniques. Pathological nodes must be = 15 mm by the short axis to be considered measurable.
* Patients aged 18 years or older, as no dosing or adverse event data are currently available on the use of afatinib in patients <18 years of age, children are excluded from this study.
* Life expectancy of at least three (3) months.
* Karnofsky performance status ≥60%
* All patients with disease technically amenable to biopsy will be asked to undergo a biopsy. Patient must agree to allow 2 biopsies of any malignant lesion that can be accessed by endoscopy or with the aid or radiology (i.e. CT guided).
* Patients who have previously provided samples at any time after trastuzumab resistance will be exempt from biopsy at the start of therapy.
* Consent to preservation of frozen and fixed samples of tumor cores for evaluation
* Able to swallow and retain oral medication.
* Negative serum HCG pregnancy test for premenopausal women of reproductive capacity and for women less than 12 months after menopause.
* Willingness to use birth control while on study.
* Asymptomatic, central nervous system metastases are permitted.

Exclusion Criteria:

* Patients receiving any concurrent anticancer therapy or investigational agents with the intention of treating esophagogastric cancer. 89Zr-trastuzumab uses as imaging agent for 89Zr-trastuzumab PET permitted.
* Prior disease progression on docetaxel or paclitaxel in metastatic setting.
* Patients who are unwilling to consent to mandatory tumor biopsy. Patients with archival tissue permitted to enroll on study per MSK Principal Investigator discretion Women who are pregnant or breast feeding.
* Concurrent radiotherapy is not permitted for disease progression on treatment on protocol (except in the context specified in section 9.0), but might be allowed for pre-existing non-target lesions with approval from the principal investigator of the trial.
* Concurrent medical conditions which may increase the risk of toxicity, including ongoing or active infection, history of significant bleeding disorder unrelated to cancer (congenital bleeding disorders, acquired bleeding disorders within one year), HIV-positive.
* Subjects with acute Hepatitis B are not eligible. Subjects with chronic hepatitis are eligible if their condition is stable and in the opinion of the investigator, if consulted, would not pose a risk to subject safety.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to study entry.
* Baseline (< 1 month before treatment) cardiac left ventricular function with resting ejection fraction of less than 50% measured by echocardiogram.
* Known pre-existing interstitial lung disease.
* Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease, malabsorption, or CTCAEGrade >2 diarrhea of any etiology.
* Unwillingness to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study.
* Active hepatitis B infection, active hepatitis C infection
* Known HIV carrier
* Known or suspected active drug or alcohol abuse. Restricted Therapies
* Additional experimental anti-cancer treatment and/or standard chemo-, immunotherapy, hormone treatment (with the exception of megestrol acetate), or concurrent radiotherapy is not allowed concomitantly with the administration of study treatment (with the exception listed in section 9.0) 89Zr-trastuzumab use as imaging agent for 89Zr-trastuzumab PET permitted. Afatinib is a substrate of P-gp and its plasma concentrations can be affected by the use of P-gp inhibitors (data on file) and it is also likely that P-gp inducers could also influence afatinib plasma concentrations.
* The use of potent P-gp inhibitors (including cyclosporine, erythromycin, ketoconazole, itraconazole, quinidine, Phenobarbital salt with quinidine, ritonavir, valspodar, verapamil) and potent P-gp inducers (including St John's wort, rifampicin) has to be avoided during treatment with afatinib. Any exemptions to this have to be discussed with the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- [Derived] Maron SB, Chatila W, Walch H, Chou JF, Ceglia N, Ptashkin R, Do RKG, Paroder V, Pandit-Taskar N, Lewis JS, Biachi De Castria T, Sabwa S, Socolow F, Feder L, Thomas J, Schulze I, Kim K, Elzein A, Bojilova V, Zatzman M, Bhanot U, Nagy RJ, Lee J, Simmons M, Segal M, Ku GY, Ilson DH, Capanu M, Hechtman JF, Merghoub T, Shah S, Schultz N, Solit DB, Janjigian YY. Determinants of Survival with Combined HER2 and PD-1 Blockade in Metastatic Esophagogastric Cancer. Clin Cancer Res. 2023 Sep 15;29(18):3633-3640. doi: 10.1158/1078-0432.CCR-22-3769. PMID 37406106
- [Derived] Sanchez-Vega F, Hechtman JF, Castel P, Ku GY, Tuvy Y, Won H, Fong CJ, Bouvier N, Nanjangud GJ, Soong J, Vakiani E, Schattner M, Kelsen DP, Lefkowitz RA, Brown K, Lacouture ME, Capanu M, Mattar M, Qeriqi B, Cecchi F, Tian Y, Hembrough T, Nagy RJ, Lanman RB, Larson SM, Pandit-Taskar N, Schoder H, Iacobuzio-Donahue CA, Ilson DH, Weber WA, Berger MF, de Stanchina E, Taylor BS, Lewis JS, Solit DB, Carrasquillo JA, Scaltriti M, Schultz N, Janjigian YY. EGFR and MET Amplifications Determine Response to HER2 Inhibition in ERBB2-Amplified Esophagogastric Cancer. Cancer Discov. 2019 Feb;9(2):199-209. doi: 10.1158/2159-8290.CD-18-0598. Epub 2018 Nov 21. PMID 30463996
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib and Paclitaxel: This is a multi-institution, open-label, non-randomized, Phase II evaluation of oral afatinib daily and intravenous paclitaxel in participants with trastuzumab refractory HER2-positive metastatic or recurrent esophagogastric adenocarcinoma.
Period: Overall Study
Arm/Group | Afatinib and Paclitaxel
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Afatinib and Paclitaxel
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 63 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Efficacy
Description: of afatinib in patients with metastatic HER2-positive esophagogastric cancer as measured by overall clinical benefit defined as response rate (ORR) = stable disease (SD) complete response (CR) or partial response (PR) at 4 months by RECIST 1.1 criteria
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib and Paclitaxel
Number analyzed (Participants) | 42
Participants
  Partial Response | 4
  Progression of Disease | 18
  Stable Disease | 12
  Not Evaluable | 8

2. Secondary Outcome: Number of Participants Evaluated for Toxicity
Description: The type, frequency, severity, timing, and relationship of each adverse event will be determined as per the NCI Common Toxicity Criteria, version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib and Paclitaxel
Number analyzed (Participants) | 42
Participants | 42

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Afatinib and Paclitaxel
All-Cause Mortality (participants affected / at risk) | 2/42
Serious Adverse Events (participants affected / at risk) | 22/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib and Paclitaxel (N=42)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 6
Acidosis (Metabolism and nutrition disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 12
Anorexia (Metabolism and nutrition disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Ataxia (Nervous system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood bilirubin increased (Investigations) | 3
Blurred vision (Eye disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Confusion (Psychiatric disorders) | 2
Conjunctivitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Death NOS (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 6
Diarrhea (Gastrointestinal disorders) | 9
Dizziness (Nervous system disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2
Gen disorders & admin site conditions Other, spec (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Hematoma (Vascular disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
INR increased (Investigations) | 3
Infections and infestations - Other (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 5
Movements involuntary (Nervous system disorders) | 1
Muscle weakness left-sided (Nervous system disorders) | 1
Muscle weakness lower limb (Nervous system disorders) | 1
Muscle weakness upper limb (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Palpitations (Cardiac disorders) | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 1
Thromboembolic event (Vascular disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib and Paclitaxel (N=42)
Diarrhea (Gastrointestinal disorders) | 38
Fatigue (General disorders) | 21
Rash acneiform (Skin and subcutaneous tissue disorders) | 18
Anemia (Blood and lymphatic system disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 12
Papulopustular rash (Skin and subcutaneous tissue disorders) | 8
Mucositis oral (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
White blood cell decreased (Investigations) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Lymphocyte count decreased (Investigations) | 4
Acute kidney injury (Renal and urinary disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Paronychia (Infections and infestations) | 3
Activated partial thromboplastin time prolonged (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 2
Gastric hemorrhage (Gastrointestinal disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Platelet count decreased (Investigations) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT01522768/Prot_SAP_000.pdf